CLINICAL TRIAL: NCT02385422
Title: The Effect of Carvedilol Vs Propranolol in Patients With Cirrhosis Related Esophagogastric Varices After Multiple Endoscopic Treatments For Secondary Prophylaxis:A Randomized Controlled Trial
Brief Title: The Effect of Carvedilol Vs Propranolol in Cirrhotic Patients With Variceal Bleeding
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Principal Investigator, Shiyao Chen, Director of department of Gastroenterology, Zhongshan Hospital, Shanghai Zhongshan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CSY-WYC-2015
Record Dates: First submitted 2015-03-04; First posted 2015-03-11 (Estimated); Last update posted 2015-03-11 (Estimated); Status verified 2015-03

CONDITIONS: Liver Cirrhosis; Esophageal and Gastric Varices; Hemorrhage
Keywords: secondary prophylaxis; Propranolol; Carvedilol; comparative effectiveness research
MeSH Terms: conditions — Liver Cirrhosis; Esophageal and Gastric Varices; Hemorrhage | interventions — Carvedilol; Propranolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Carvedilol (Experimental): Carvedilol，6.25mg-25mg/d,oral,6 months
  Interventions: Drug: Carvedilol
- Propranolol (Active Comparator): Propranolol,30mg-160mg/d,oral,6 months
  Interventions: Drug: Propranolol

INTERVENTIONS:
Drug: Carvedilol — Carvedilol is started at a dose of 6.25mg/d, and titrated to a maximum dose of 25mg/d. Doses are increased every 2-3 days until ABPsys is not less than 90 mm Hg and HR is not less than 55 bpm.
  Other Names: JinLuo
  Arms: Carvedilol
Drug: Propranolol — Patients receiving propranolol start at a dose of 30 mg/d and the dose will be increased to a maximum dose of 160 mg/d.Doses are increased every 2-3 days until ABPsys is not less than 90 mm Hg and HR is not less than 55 bpm.
  Other Names: XinDeAn
  Arms: Propranolol

SUMMARY:
To compare the efficacy and safety of Carvedilol and Propranolol in patients with cirrhosis-related esophagogastric varices after multiple endoscopic treatments for secondary prophylaxis.

DETAILED DESCRIPTION:
The study is a randomized controlled trial. Patients randomly enter into two treatment groups: 1)the Carvedilol group and 2)the Propranolol group. Treatment allocation is by block randomization, with an equal number for Carvedilol and Propranolol. The results are concealed in opaque envelopes. The dose of non-selective β-blocker(NSBB) is titrated according to systolic arterial blood pressure (ABPsys) and heart rate (HR). Doses are increased every 2-3 days until ABPsys is not less than 90 mm Hg and HR is not less than 55 bpm. Carvedilol is started at a dose of 6.25mg/d, and titrated to a maximum dose of 25mg/d. Patients receiving propranolol start at a dose of 30 mg/day and the dose will be increased to a maximum dose of 160 mg/day. Patients will be followed up with telephone calls every 2 months. After taking these 2 drugs for 6 months, patients come for clinic visits, receiving laboratory tests and endoscopic examinations, and events of primary and secondary outcomes will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* age between 18-70 years old;
* cirrhotic patients referred to Zhongshan Hospital with esophagogastric varices confirmed by endoscopy;
* history of variceal bleeding; at least 3 times of endoscopic treatment;
* with 1) mild esophageal varices;2) gastric varices with a diameter less than 5mm; or 3) variceal eradication at the time of recruiting.

Exclusion Criteria:

Patients are excluded when they have

* episodes of variceal bleeding after the last endoscopic treatment;
* diagnosis of hepatic cellular carcinoma;
* severe systemic diseases;
* refractory ascites;
* contraindication to Carvedilol or Propranolol, such as: asthma, chronic obstructive pulmonary disease, allergic rhinitis, New York Heart Association IV chronic heart failure, atrioventricular blockade, severe bradycardia(HR<50bpm), sick sinus syndrome, cardiogenic shock, severe hypotension(ABPsys<85mmHg);
* previous and continued use of β-blockers;
* Child -Pugh Class C.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2015-03; Primary Completion 2017-06 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Endoscopic Retreatment | 6 months
  Patients will receive an endoscopic examination after they have been followed up for 6 months, and if they have recurrence of varices or deterioration of varices,they are considered to be in need of endoscopic retreatment.

SECONDARY OUTCOMES:
Rebleeding rate | 6 months
  We observe the variceal rebleeding events during 6 months.
Mortality rate | 6 months
  We observe the mortality events during 6 months due to variceal bleeding, hepatic encephalopathy, liver failure, hepatic cellular carcinoma, hepatic-renal syndrome and spontaneous bacterial peritonitis.
Adverse events | 6 months
  We observe any severe adverse events caused by drug treatment,including palpitation,bronchospasm,syncope,dizziness,hypotension,ascites,edema,bradycardia.

CONTACTS AND LOCATIONS:
Overall Officials: Shiyao Chen, Professor, Study Director — Shanghai Zhongshan Hospital
Locations (1):
- Shanghai Zhongshan Hospital, Shanghai, Shanghai Municipality, China